CLINICAL TRIAL: NCT02015078
Title: Black Family Eating Behaviors Study
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Collaborators: Duke University (Other); National Cancer Institute (NCI) (NIH); University of North Carolina (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914014; 14-HG-N014
Record Dates: First submitted 2013-12-14; First posted 2013-12-19 (Estimated); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Cancer; Obesity
Keywords: African American; Eating Behavior Phenotypes; Obesity; Natural History
MeSH Terms: conditions — Neoplasms; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- African Americans: Targets are family members attending African American family reunions.

SUMMARY:
Despite broad awareness of the role that diet plays in increasing obesity risk, adherence to public health recommendations for maintaining healthy eating is low. Insights gained from weight loss intervention trials find that trial participants report difficulty in restricting calories, dissatisfaction with the pace of weight loss, inability to control eating, low palatability of recommended foods and strong food cravings. Indeed, recent systematic reviews provide empirical support that these subjective experiences that trial participants describe likely represent eating-related traits or phenotypes . While amassing evidence supports individual variation in these eating-related traits, to date there has been no systematic effort to characterize robust eating-related phenotypes. Proposed is a Sub-study initially planned to be piggy-backed on a planned Study being conducted by investigators at the University of North Carolina (UNC-- Linnan, Dilworth- Anderson & Evans). The UNC Parent Study was a feasibility study using community-based participatory research (CBPR) approaches to explore possible intervention strategies aimed to reduce the burden of chronic disease and cancer among African American families. The NHGRI-led eating behavior Sub-study is proposed to be integrated with the UNC Parent Study (hereafter referred to as Phase 1). The additional aims of the Sub-study (hereafter referred to as Phase 2) are to gain understanding of whether we can characterize clusters of eating-related behaviors that may be associated with adherence to weight management and weight outcomes. This current protocol lays out the specific qualitative activities planned for Phase 1 which include conducting structured interviews with Black Family Reunion organizers (N=8) and a sample of reunion participants (N=40). We also describe the larger quantitative survey proposed for Phase 2. Pending the feasibility of the sub-study with the African-American community, we will collect information on eating-related behaviors in a large sample of individuals (N=350). If the initial assessments (Phase1) prove that this is not a viable study to be conducted in that setting, we will consider other population groups and other settings.

We are also considering Phase 3 activities if we identify clusters of eating-related phenotypes within individuals. Amended IRB applications will be submitted prior to launching Phase 3.

DETAILED DESCRIPTION:
Despite broad awareness of the role that diet plays in increasing obesity risk, adherence to public health recommendations for maintaining healthy eating is low. Insights gained from weight loss intervention trials find that trial participants report difficulty in restricting calories, dissatisfaction with the pace of weight loss, inability to control eating, low palatability of recommended foods and strong food cravings. Indeed, recent systematic reviews provide empirical support that these subjective experiences that trial participants describe likely represent eating-related traits or phenotypes . While amassing evidence supports individual variation in these eating-related traits, to date there has been no systematic effort to characterize robust eating-related phenotypes. Proposed is a Sub-study initially planned to be piggy-backed on a planned Study being conducted by investigators at the University of North Carolina (UNC-- Linnan, Dilworth- Anderson & Evans). The UNC Parent Study was a feasibility study using community-based participatory research (CBPR) approaches to explore possible intervention strategies aimed to reduce the burden of chronic disease and cancer among African American families. The NHGRI-led eating behavior Sub-study is proposed to be integrated with the UNC Parent Study (hereafter referred to as Phase 1). The additional aims of the Sub-study (hereafter referred to as Phase 2) are to gain understanding of whether we can characterize clusters of eating-related behaviors that may be associated with adherence to weight management and weight outcomes. This current protocol lays out the specific qualitative activities planned for Phase 1 which include conducting structured interviews with Black Family Reunion organizers (N=8) and a sample of reunion participants (N=40). We also describe the larger quantitative survey proposed for Phase 2. Pending the feasibility of the sub-study with the African-American community, we will collect information on eating-related behaviors in a large sample of individuals (N=350). If the initial assessments (Phase1) prove that this is not a viable study to be conducted in that setting, we will consider other population groups and other settings.

We are also considering Phase 3 activities if we identify clusters of eating-related phenotypes within individuals. Amended IRB applications will be submitted prior to launching Phase 3.

ELIGIBILITY:
* INCLUSION
* For Phase 1 of the study, targets are family members attending African American family reunions. Therefore, the eligibility to participate will be: age 18 or older; not currently pregnant; attending the targeted family reunion.
* For Phase 2 of the study, the population for the study are adults (18 to 70 years-old), with the capability to read English. As this is a feasibility and exploration study, the recruitment is intended to be broad and to include various populations and profiles.

EXCLUSION

-Pregnant women will be excluded from participation in the study due to the focus on eating behaviors and weight.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Targets are family members attending African American family reunions.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2013-12-14; Primary Completion 2015-04-15 (Actual); Study Completion 2015-06-22 (Actual)

PRIMARY OUTCOMES:
Phase 3 | Completed
  To assess whether the occurrence of robust eating- related behavior clusters differ significantly between blood relatives and non-blood relatives (i.e., spouses and unrelated kin).
Phase 2 | Completed
  To assess whether robust phenotypes of eating-related behaviors (e.g., appetite for palatable foods, disinhibition, pickiness, and new food phobia) can be characterized.
Phase 1 | Completed
  To assess the feasibility of:(a)recruiting African American family reunion-organizers and participants to take part in a health promotion and genetics- related research study. (b)administering survey assessments to assess individual s and kindreds (blood and nonblood relatives ) interest in learning about eating-related (ER) behaviors and weight outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Persky, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Akter SM, Roy SK, Thakur SK, Sultana M, Khatun W, Rahman R, Saliheen SS, Alam N. Effects of third trimester counseling on pregnancy weight gain, birthweight, and breastfeeding among urban poor women in Bangladesh. Food Nutr Bull. 2012 Sep;33(3):194-201. doi: 10.1177/156482651203300304. PMID 23156122
- [Background] Appelhans BM, Woolf K, Pagoto SL, Schneider KL, Whited MC, Liebman R. Inhibiting food reward: delay discounting, food reward sensitivity, and palatable food intake in overweight and obese women. Obesity (Silver Spring). 2011 Nov;19(11):2175-82. doi: 10.1038/oby.2011.57. Epub 2011 Apr 7. PMID 21475139
- [Background] Baranowski T, Baranowski JC, Watson KB, Jago R, Islam N, Beltran A, Martin SJ, Nguyen N, Tepper BJ. 6-n-propylthiouracil taster status not related to reported cruciferous vegetable intake among ethnically diverse children. Nutr Res. 2011 Aug;31(8):594-600. doi: 10.1016/j.nutres.2011.07.004. Epub 2011 Aug 5. PMID 21925344
- [Derived] Persky S, Bouhlal S, Goldring MR, McBride CM. Beliefs about genetic influences on eating behaviors: Characteristics and associations with weight management confidence. Eat Behav. 2017 Aug;26:93-98. doi: 10.1016/j.eatbeh.2017.02.003. Epub 2017 Feb 9. PMID 28199907